CLINICAL TRIAL: NCT03573089
Title: An Investigator-initiated, International, Multi-centre, Prospective, Randomized, Open-label, Parallel-group, Superiority, and Pragmatic Large Simple Trial (LST) to Determine Whether the Currently Recommended Strategy of Intensive Reduction of Serum Phosphate Concentration Towards the Normal Level Results in Significant Patient-centred Benefits in End-stage Kidney Disease (ESKD) Patients Receiving Dialysis.
Brief Title: Pragmatic Randomised Trial of High Or Standard PHosphAte Targets in End-stage Kidney Disease (PHOSPHATE)
Acronym: PHOSPHATE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Queensland (Other)
Collaborators: National Health and Medical Research Council, Australia (Other); Applied Health Research Centre (Other); Cambridge University Hospitals NHS Foundation Trust (Other); University of Otago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AKTN 17.02
Record Dates: First submitted 2018-05-20; First posted 2018-06-29 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2024-09

CONDITIONS: Kidney Failure, Chronic; Hyperphosphatemia
Keywords: Renal dialysis; Randomised controlled trial; Bone markers; Cardiovascular risk factors; Phosphate lowering agent; End stage kidney disease; Hyperphosphatemia
MeSH Terms: conditions — Kidney Failure, Chronic; Hyperphosphatemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Liberal phosphate target (Active Comparator): Liberal serum phosphate target of 2.0 to 2.5 mmol/L.
  Interventions: Drug: Liberal phosphate target
- Intensive phosphate target (Experimental): Intensive serum phosphate target of ≤1.50 mmol/L.
  Interventions: Drug: Intensive phosphate target

INTERVENTIONS:
Drug: Liberal phosphate target — All phosphate-lowering medications in use at baseline will be discontinued. Phosphate-lowering medications will be prescribed only if serum phosphate concentration exceeds 2.50 mmol/L. The choice and dosages of phosphate-lowering medications will be at the discretion of treating physicians and/or participants.
  Arms: Liberal phosphate target
Drug: Intensive phosphate target — This will be achieved by prescribing phosphate-lowering medications aimed to intensively lower serum phosphate concentration towards normal level (≤1.50 mmol/L). The choice and dosages of phosphate-lowering medications will be at the discretion of treating physicians and/or participants.
  Arms: Intensive phosphate target

SUMMARY:
During end-stage kidney disease, clinical guidelines suggest reducing elevated phosphate levels in the blood. However, the effect of lowering blood phosphate levels on important patient-centred outcomes has never been tested. This trial will evaluate whether compared to high levels, lowering blood phosphate levels would reduce death or major events due to heart disease, improve physical health, and be cost-effective.

DETAILED DESCRIPTION:
Hyperphosphataemia is highly prevalent in patients with end-stage kidney disease (ESKD) and associated with increased mortality risk. The Clinical Practice Guidelines suggest lowering elevated phosphate levels towards the normal range (level 2C suggestion). However, trial data demonstrating that treatments that lower serum phosphate will improve patient-centred outcomes are lacking.

The primary objective is to test the hypothesis that compared to a liberal serum phosphate concentration target of 2.0 to 2.5 mmol/L, intensive lowering of serum phosphate towards the normal level (≤1.50 mmol/L) with phosphate binders reduces the risk of fatal or non-fatal major cardiovascular events in ESKD patients receiving dialysis. The secondary objectives are to test the hypothesis that intensive lowering of serum phosphate towards the normal level with phosphate binders would improve physical health, fatigue, health-related quality of life, patient satisfaction, and pruritus; and be cost-effective.

In this pragmatic, multinational, randomised controlled large simple trial, a total of 3600 adult ESKD patients receiving dialysis will be randomised either to intensive (≤1.50 mmol/L) or liberalized (2.0-2.5 mmol/L) serum phosphate target. The choice and dose of phosphate binders will be at the treating physician's discretion and local practice to achieve and maintain serum phosphate concentration within the required target range according to randomisation. The primary endpoint is the composite endpoint of cardiovascular death, non-fatal major cardiovascular or peripheral arterial events. The secondary outcome measures will be individual components of the primary composite endpoint, all-cause death, and utility-based quality of life EQ5D-5L.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥45 years, or Age ≥18 years with diabetes,
2. ESKD on haemodialysis or peritoneal dialysis, for at least 3 months,
3. Currently prescribed at least one phosphate-lowering medication at any dose
4. Able to provide informed consent

Exclusion Criteria:

1. Elective kidney transplantation scheduled,
2. Concomitant major illness / comorbidity that may result in death in the next 6 months in the view of the treating physician,
3. Participation in an interventional study that is likely to affect serum phosphate concentration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3600 (Estimated)
Dates: Start 2019-12-10 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to a composite endpoint of cardiovascular death or non-fatal major cardiovascular event | 5 years
  Time to a composite endpoint of cardiovascular death, non-fatal myocardial infarction or coronary revascularization, stroke, or peripheral arterial event.

SECONDARY OUTCOMES:
Time to individual components of the primary composite endpoint, | 5 years
Time to all-cause death | 5 years
Utility-based quality of life EQ5D-5L | 5 years
  EQ5D-5L will be used to assess patient self-reported quality of life measures.

OTHER OUTCOMES:
Differences in the serum concentrations of phosphate, PTH, calcium, alkaline phosphatase and albumin | Time Frame: 5 years
Phosphate-lowering medication usage | 5 years
Phosphate-lowering medication self-reported adherence | 5 years
Proportion of patients requiring parathyroidectomy | 5 years
Proportion of patients developing calciphylaxis | 5 years
Gastrointestinal Symptom Rating Scale | 5 years
  The Gastrointestinal Symptom Rating Scale (GSRS) is a 15-item instrument designed to assess the symptoms associated with common GI disorders. It has five subscales (reflux, diarrhea, constipation, abdominal pain and indigestion). Subscale scores range from 1-7 and higher scores represent higher symptom burden i.e. more discomfort.
Itch/pruritus visual analog scale | 5 years
  The Pruritis 5-D scale contains five domains: duration, degree, direction, disability and distribution. The scores of each of the five domains are achieved separately and then summed together to obtain a total 5-D score. 5-D scores can potentially range between 5 (no pruritus) and 25 (most severe pruritus).
Cost-effectiveness analysis: | 5 years
  Difference in the incremental cost per Quality Adjusted Life Years gained

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Badve, Principal Investigator — The University of Queensland; Ron Wald, Principal Investigator — St Michael's Hospital; Rona Smith, Principal Investigator — University of Cambridge; Suetonia Green, Principal Investigator — University of Otago; Patrick Mark, Principal Investigator — University of Glasgow; Rathika Krishnasamy, Principal Investigator — The University of Queensland; Michael Walsh, Principal Investigator — Hamilton Centre for Kidney Research
Locations (115):
- Australia (23):
  - Royal Prince Alfred Hosptial, Camperdown, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - Royal North Shore Hospital, Saint Leonards, New South Wales
  - Western Sydney Renal Service, Westmead, New South Wales
  - Wollongong Hospital, Wollongong, New South Wales
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Bundaberg Hospital, Bundaberg, Queensland
  - Cairns Hospital, Cairns, Queensland
  - Fraser Coast Renal Service, Hervey Bay, Queensland
  - Mackay Hospital, Mackay, Queensland
  - Logan Hospital, Meadowbrook, Queensland
  - Gold Coast University Hospital, Southport, Queensland
  - Townsville University Hospital, Townsville, Queensland
  - Central and Northern Adelaide Renal and Transplant Service, Adelaide, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
  - Austin Health, Heidelberg, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
  - St Vincent's Hospital Melbourne, Melbourne, Victoria
  - Latrobe Regional Hospital, Traralgon, Victoria
  - Armadale Hospital, Armadale, Washington
- Brazil (5):
  - BRA Santa Casa de Misericórdia de Ponta Grossa, Ponta Grossa, Paraná
  - Sociedade Hospitalar Angelina Caron, Campina Grande, Paraíba
  - Hospital de Clinicas Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Fundacao Felice Rosso - Hospital Felicio Rocho, Barro Preto
  - Hospital Alemao Oswaldo Cruz, São Paulo
- Canada (30):
  - Foothills Hospital/ U of Calgary, Calgary, Alberta
  - Alberta Health Services, Edmonton, Alberta
  - St. Paul's Hospital, Vancouver, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - Dalhousie University, Halifax, Nova Scotia
  - Queen's University, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - Oakville Trafalgar Memorial Hospital, Oakville, Ontario
  - Orillia Soldier's Memorial Hospital, Orillia, Ontario
  - Lakeridge Health, Oshawa, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Mackenzie Health, Richmond Hill, Ontario
  - Scarborough Hospital Network, Scarborough Village, Ontario
  - St Michael's Hospital, Toronto, Ontario
  - University Health Network - University of Toronto, Toronto, Ontario
  - St. Joseph's Healthcare Hamilton, Toronto, Ontario
  - St. Joseph's Healthcare Toronto, Toronto, Ontario
  - The Charles Lemoyne Hospital, Longueuil, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - Hopital Maisonneuve Rosemont, Montreal, Quebec
  - CHUM, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - Sacre Coeur Hospital, Montreal, Quebec
  - CHU de Quebec Universite Laval, Québec, Quebec
  - Centre hospitalier universitaire de Sherbrooke (CHUS), Sherbrooke, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec
  - Red Deer Hospital;, Red Deer
  - Humber River Hospital, Toronto
  - Michael Garron Hospital, Toronto
  - Trillium Health Partners, Toronto
- AURA Paris Plaisance, Paris, France
- Israel (4):
  - Hadassah University, Jerusalem
  - Shaare Zedek Medical Centre, Jerusalem
  - Meir Hospital, Kfar Saba
  - Sheba Hospital, Ramat Gan
- New Zealand (8):
  - Auckland City Hospital, Auckland
  - Christchurch Hospital, Christchurch
  - Dunedin Hospital, Dunedin
  - Waikato DHB, Hamilton
  - Hawkes Bay Hospital, Hastings
  - Middlemore Hospital, Otahuhu
  - Waitematā Hospital, Takapuna
  - Northland DHB, Whangarei
- Ramathibodi Hospital, Bangkok, Khet Ratchathewi, Thailand
- United Kingdom (43):
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge, Cambridgeshire
  - University Hospitals Plymouth NHS Trust, Plymouth, Devon
  - Dorset County Hospital NHS Foundation Trust, Dorchester, Dorset
  - South Tyneside And Sunderland NHS Foundation Trust, Sunderland, Durham
  - East and North Hertfordshire NHS Trust, Stevenage, Hertfordshire
  - East Kent Hospitals University NHS Foundation Trust, Canterbury, Kent
  - NHS Greater Glasgow and Clyde, Glasgow, Kent
  - James Paget University Hospitals NHS Foundation Trust, Great Yarmouth, Norfolk
  - NHS Lanarkshire, Airdrie, North Lanarkshire
  - South Tees Hospitals NHS Foundation Trust, Middlesbrough, North Yorkshire
  - York and Scarborough Teaching Hospitals NHS Foundation Trust, York, North Yorkshire
  - Nottingham University Hospitals NHS Trust, Nottingham, Nottinghamshire
  - NHS Highland, Inverness, Scotland
  - Shrewsbury and Telford Hospital NHS Trust, Shrewsbury, Shropshire
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, South Yorkshire
  - University Hospital of North Midlands NHS Trust, Stoke-on-Trent, Staffordshire
  - West Suffolk Hospital, Bury St Edmunds, Suffolk
  - University Hospitals Sussex NHS Foundation Trust, Brighton, Sussex
  - Bradford Teaching Hospital NHS Foundation Trust, Bradford, West Yorkshire
  - Wirral University Teaching Hospital NHS Foundation Trust, Birkenhead, Wirral
  - University Hospital Birmingham NHS foundation Trust, Birmingham
  - Cardiff and Wales University Local Health Board, Cardiff
  - North Cumbria Integrated Care NHS Foundation Trust, Carlisle
  - Epsom and St Helier University Hospitals NHS Trust, Carshalton
  - Gloucestershire Hospital NHS Foundation Trust, Cheltenham
  - University Hospitals Coventry & Warwickshire, Coventry
  - University Hospitals of Derby and Burton, Derby
  - Doncaster and Bassetlaw Teaching Hospitals NHS Foundation Trust, Doncaster
  - The Dudley Group NHS Foundation Trust, Dudley
  - Royal Devon and Exeter NHS Foundation Trust, Exeter
  - Hull University Teaching Hospital NHS Trust, Hull
  - Ipswich Hospital (East Suffolk & North Essex Foundation Trust), Ipswich
  - University Hospitals Of Leicester NHS Trust, Leicester
  - Royal Liverpool University Hospitals, Liverpool
  - University Hospital Aintree, Liverpool
  - Guy's and St Thomas' NHS Foundation Trust, London
  - King's College Hospital NHS Foundation Trust, London
  - St George's University Hospitals NHS Foundation Trust, London
  - Manchester University NHS Foundation Trust, Manchester
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne
  - Royal Berkshire NHS Foundation Trust, Reading
  - Mid and South Essex NHS Foundation Trust, Southend-on-Sea
  - The Royal Wolverhampton NHS Trust, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the primary publication, after deidentification (text, tables, figures and appendices) will be available for individual participant data meta-analysis.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 2 years and ending 5 years following main publication. Proposals may be submitted up to 5 years following article publication. After 5 years, the data will be available in our University's data warehouse but without investigator support other than deposited metadata.
Access Criteria: An independent review board will assess proposals based on the following criteria: sound science, benefit-risk balancing and research team expertise.

REFERENCES:
- [Derived] Edmonston D, Isakova T, Dember LM, Waymyers S, Andersen D, Chan KE, Chakraborty H, Wolf M. Higher versus Lower Phosphate Targets for Patients Undergoing In-Center Hemodialysis: A Randomized Controlled Trial. J Am Soc Nephrol. 2025 Dec 1;36(12):2445-2455. doi: 10.1681/ASN.0000000765. Epub 2025 Jul 10. PMID 40638247
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086
- [Derived] Fajol A, Faul C. The Pathologic Actions of Phosphate in CKD. Kidney360. 2025 Apr 17;6(6):1040-1049. doi: 10.34067/KID.0000000820. PMID 40241437
- [Derived] Fernandez L, Klein J. Vascular Calcification and CKD: Challenges, Emerging Targets, and Future Perspectives. Clin J Am Soc Nephrol. 2025 Nov 1;20(11):1630-1633. doi: 10.2215/CJN.0000000733. Epub 2025 Apr 16. No abstract available. PMID 40238244
- [Derived] Edmonston D. Tight Phosphate Control in ESKD Patients Is Warranted: CON. Kidney360. 2024 Dec 13;6(6):895-897. doi: 10.34067/KID.0000000000000401. No abstract available. PMID 39671553
- See also: Australasian Kidney Trials Network Website — http://aktn.org.au/